CLINICAL TRIAL: NCT07351903
Title: The Single-arm Open-label Clinical Study Evaluating the Use of GK01 Cell Injection in Combination With or Without Chemotherapy for the Adjuvant Treatment of Solid Tumors
Brief Title: A Single-arm, Open-label Study of GK01 in Combination With or Without Chemotherapy for the Adjuvant Treatment of Solid Tumors
Acronym: GUARDIAN-02
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Beijing Geekgene Technology Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GUARDIAN-02
Record Dates: First submitted 2026-01-11; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GK01 injection (Experimental): Autologous tumor-reactive T cells injection
  Interventions: Drug: GK01 Injection

INTERVENTIONS:
Drug: GK01 Injection — Autologous tumor-reactive T cells injection

SUMMARY:
This study is an open-label, single-arm clinical trial to evaluate the safety, pharmacokinetics, and preliminary efficacy of GK01 in patients with advanced solid tumors.

ELIGIBILITY:
* Ability to understand and sign a written informed consent document.
* At the date of signing ICF, 18 ~70 years old, male or female.
* Patients with solid tumors confirmed by histopathology (including but not limited to pancreatic cancer, cholangiocarcinoma, gastric cancer, etc.) who are judged by investigator to be capable of undergoing radical total resection of the primary tumor for the purpose of cure.
* No treatment for the primary tumor was received before surgical resection (no induction therapy or recurrent disease).
* The expected survival time is more than 12 weeks;.
* ECOG 0-1 points.

Exclusion Criteria:

* Inoperable or metastatic (Stage IV) solid tumors.
* Central nervous system (CNS) metastasis, leptomeningeal disease, or metastatic spinal cord compression; or a history of CNS disorders, including but not limited to epilepsy, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, etc.
* History of bone marrow or solid organ transplantation.
* History of other primary malignancies within 5 years prior to study treatment
* Hepatitis B surface antigen (HBsAg) positivity; With negative HBsAg but positive hepatitis B core antibody (HBcAb) ,and if peripheral blood hepatitis B virus (HBV) DNA positive; Hepatitis C virus (HCV) antibody positive and HCV RNA positive; Human immunodeficiency virus (HIV) antibody positive; Cytomegalovirus (CMV) DNA positive; Both Treponema pallidum-specific and non-specific antibody tests are positive.
* Allergy to any components of the drugs planned.
* Previous radiotherapy within 28 days before signing the ICF.
* History of active tuberculosis infection within 1 year before screening.
* Concurrent or previous history of interstitial lung disease or interstitial pneumonia; presence of chronic lung disease or other respiratory conditions that significantly impair lung function.
* Diagnosis of active autoimmune disease or a history of autoimmune disease that may recur (e.g., systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vasculitis, psoriasis, etc.), or at risk of such conditions.
* Investigator-assessed clinically significant thyroid dysfunction.
* Cardiovascular diseases with clinical significance.
* No contraindications to curative resection of the primary tumor.
* Attenuated or inactivated vaccines within 28 days before signing the I form, or planned administration of such vaccines during the screening period.
* Comorbidities or other conditions are likely to affect protocol compliance or suitability for participation in this study.
* Female subjects who are pregnant or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2028-10-15 (Estimated); Study Completion 2029-02-14 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 2 years
  The incidence and severity, and correlation of AEs (Adverse Events) and SAEs (Serious Adverse Events).

SECONDARY OUTCOMES:
PK | 2 years
  Levels of T-cell Receptor copies
Recurrence free survival(RFS) | 2 years
  RFS will will be assessed from radical surgery to death of any cause (evaluated according to the RECIST criteria).
Overall survival (OS ) | 2 years
  OS will be assessed from the first GK01 infusion to death from any cause (Assessed based on RECIST criteria)
Patient Quality of Life | 2 years
  EORTC(European Organisation for Research and Treatment of Cancer) QLG (Quality of Life Group)Core Questionnaire (EORTC QLQ-C30)
PD marker | 2 years
  Concentration levels of serum cytokines, tumor markers and other related markers.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Cancer Hospital Airport Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No